CLINICAL TRIAL: NCT05774301
Title: Effect of a Structured Simulation-based Training on Oncology Nurses' Performance Regarding Port A Cath Device.
Brief Title: Structured Training on Oncology Nurses' Performance Related Port A Cath Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Abubakr Mohamed Salama, Assistant Professor, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: training on port A cath device
Record Dates: First submitted 2023-03-02; First posted 2023-03-17 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Port a Cath
Keywords: simulated training, oncology nurses, port a cath device

STUDY DESIGN:
Intervention Model Description: pre- and post-test
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurses (Experimental): A simulation-based training will be done for all nurses
  Interventions: Behavioral: simulation-based training

INTERVENTIONS:
Behavioral: simulation-based training — the training will include a theoretical & practical parts

SUMMARY:
evaluate the effect of structured simulation-based training on oncology nurses' performance regarding port A cath device.

DETAILED DESCRIPTION:
All oncology nurses who are expected to deal with port a-cath device will be recruited in the study pre test will introduced first, then simulated based training will be placed related to port a-cath device care after that , post test will be done immediately and 3 months later to measure nurses knowledge and practice level

ELIGIBILITY:
Inclusion Criteria:

* Oncology nurses who are providing direct care for patients with port a-cath device

Exclusion Criteria:

* Participants who will not be able to complete the questionnaire

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
change in oncology nurses' knowledge and practice regarding port a-cath device care | 3 months
  The researchers will provide a structured questionnaire based on reviewing related literatures called "Port a-Cath Nurses Knowledge questionnaire", it will consist of closed-ended questions to assess Nurses Knowledge And they will assess Nurses Practice level by using the preprepared Port a-Cath Nurses observational checklist.
  They will be used three times: before, immediately after training and 3 months post training

CONTACTS AND LOCATIONS:
Overall Officials: faculty of Nursing, Study Chair — Mansoura University
Locations (1):
- Heba Abubakr Salama, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No